CLINICAL TRIAL: NCT06814392
Title: Renal and Urinary Manifestations of Chronic Inflammatory Bowel Diseases: Prevalence, Risk Factors, and Prevention of Kidney Diseases in Patients With IBD, and Management of Transplant Patients.
Brief Title: Renal and Urinary Manifestations of Chronic Inflammatory Bowel Diseases.
Status: Active, not recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: I-RENE
Record Dates: First submitted 2025-01-10; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2024-10

CONDITIONS: IBD - Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The association between IBD and kidney diseases is more common than previously thought. However, the data is limited and comes from studies with small sample sizes. The proposed study aims to investigate this association in a large population of patients with IBD, assessing risk factors and potential changes in the therapeutic approach to minimize the risk of kidney damage.

The primary objective of this study is to characterize the association between IBD and kidney diseases, as well as the progression of intestinal disease and kidney function in patients who have undergone transplantation.

The study is monocentric, observational, and both retrospective and prospective.

DETAILED DESCRIPTION:
All patients who agree to participate in the study and sign the informed consent will be asked to allow the collection of their clinical data for database compilation. Retrospective data will be evaluated and collected from the medical records of all patients with Chronic Inflammatory Bowel Diseases followed at the SSD Chronic Inflammatory Bowel Diseases center. For patients with a diagnosis of kidney disease still affiliated with the center, prospective data collection will occur for a period of 3 years from enrollment in the study. No additional study-specific analyses or procedures are planned.

* Sample Size Approximately 1500 patients with Chronic Inflammatory Bowel Diseases are expected to be enrolled.
* Statistical Analysis All analyses will be performed using Stata 13.0 for Windows. The characteristics of the enrolled and observed patients will be summarized using descriptive statistics. All variables will be summarized with descriptive statistical analyses. For qualitative variables: relative frequency and 95% confidence intervals; for quantitative variables: mean, standard deviation, and percentiles. To detect possible associations between observed qualitative characteristics, Pearson's Chi-square test will be used, along with Yates' continuity correction or Fisher's exact test. Analysis of variance (ANOVA) or analysis of covariance (ANCOVA) will be used for quantitative variables.

Statistical analysis will be conducted using the Stats package. Differences between groups will be evaluated with Student's t-test and uni- and multivariate analyses to identify risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age ≥ 18 years
* Diagnosis of Crohn's Disease or Ulcerative Colitis

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Chronic Inflammatory Bowel Diseases who have been followed at the SSD Chronic Inflammatory Bowel Diseases center. For patients with a diagnosis of kidney disease still affiliated with the center, data collection will be conducted prospectively for a period of 3 years from enrollment in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2021-10-20 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary objective of this study is to characterize the association between IBD and kidney diseases, as well as the progression of intestinal disease and kidney function in patients who have undergone transplantation. | From enrollment to the end of study at 3 years
  Assess the prevalence of kidney diseases in a large population of patients with IBD; Evaluate the course of IBD and the outcomes of kidney transplantation; Identify potential risk factors for the development of kidney diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Rizzello, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy